CLINICAL TRIAL: NCT00596765
Title: Phase 2 Study of Neuropsychological Therapy for Patients With Acquired Brain Injury Focusing on the Role of Psychosocial Adjustment Using a Cognitive Behavioral Approach
Brief Title: Neuropsychological Cognitive Behavioral Therapy for Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr. Winfried Rief, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuroPsy_Ex2007
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Brain Injury
Keywords: Brain Injury; Neuropsychology; Cognitive Behavioral Therapy; Neuropsychological Rehabilitation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Neuropsychological cognitive behavioral psychotherapy for patients with acquired brain injury consists of 25 weekly 1-hr sessions of individualized outpatient treatment. The therapeutical intervention is modularised, patients are assigned to specific interventional modules according to the results of cognitive testing and interviews. Modules concern on the one hand the treatment of deficits in attention, memory, and executive functions. On the other hand psychosocial adjustment to chronic illness is addressed through modules that concern the development of a positive self-concept, the adjustment of life-goals and coping with negative affect (e.g. depressive symptoms, irritability, guilt).
  Interventions: Behavioral: Neuropsychological Cognitive Behavioral Therapy
- 2 (Other): Waiting list: Patients are randomly assigned to one of two existing groups after completion of the first session of various neuropsychological tests and interviews.
  Patients assigned to the experimental group receive therapy immediately after completing the first session of various neuropsychological tests and interviews. Patients randomized to the waiting list receive the treatment as specified above after waiting for 5 month.
  Interventions: Behavioral: Neuropsychological Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Neuropsychological Cognitive Behavioral Therapy — Neuropsychological Cognitive Behavioral Therapy encompasses 2 foci: First emphasis is on neuropsychological compensatory strategies for the treatment of deficits in attention, memory, and executive functions. Secondly, cognitive behavioral intervention techniques are employed to support the patient in the process of coping with chronic illness: i.e. improve regulation of negative affect, diversify the impaired self-concept after acquired brain injury, and adjust important life-goals to changed circumstances.

SUMMARY:
Acquired brain injury can result in impaired everyday functioning as well as psychosocial problems, including depressive symptoms, irritability, or negative self-concept. The purpose of this study is to determine whether a combination of neuropsychological and cognitive behavioral therapy is effective in the treatment of these sequelae.

DETAILED DESCRIPTION:
Acquired brain injury (ABI) commonly results in persistent cognitive, emotional and motivational problems. About 50% of patients involved develop psychiatric illness, most likely in the first year following ABI, which is associated with reduced psychosocial functioning and less favorable rehabilitation outcome. Treatment of these complex conditions requires a combination of neuropsychological and psychotherapeutic intervention techniques.

This study aims at evaluating a combination of neuropsychological intervention methods, which include developing and using compensation strategies for cognitive impairments (attention, memory and executive functions), and psychotherapeutic intervention focusing on emotion regulation, developing positive self-concepts and adjustment of life-goals. These therapeutic interventions are modularized and patients are assigned to intervention modules according to results of objective neuropsychological testing and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered an acquired brain injury after the age of 14, such as traumatic brain injury, neoplasm (after surgery), toxic brain damage, or brain damages through inflammatory diseases
* Being at least 3 months post injury
* Being German-speaking
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* Suffering from recurrent, degenerative, or progressive neurological diseases (e.g. multiple sclerosis, dementia, Chorea Huntington)
* Current or past psychosis or bipolar disorder
* Current or past diagnosis of substance dependency
* History of mental retardation
* Currently in psychotherapy
* Severe lateralized disorder (e.g. aphasia, neglect)
* Lacking minimum basic skills for attending therapy (e.g. not orientated to person, place, time, and events; unable to sustain attention for an hour-long session; cannot state cognitive strengths and weaknesses; cannot state areas in everyday functioning that are impaired due to the acquired brain injury)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-09; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Psychosocial Adjustment/ Everyday Functioning as a composite score of SCL-90-R and AFIB | Pre-/ Post-Design, including 3 ponts of measurement: at the beginning of therapy/ waiting period; immediately after completion of therapy/ waiting period; catamnestic measurement 6 months later

SECONDARY OUTCOMES:
Quality of Life (Qolibri, Seiqol, SWLS) | Pre-/ Post-Design, including 3 points of measurement: at the beginning of therapy/ waiting period; immediately after completion of therapy/ waiting period; catamnestic measurement 6 months later
Self-concept/ Life Goals (HISDS II; GOALS; RSES-REV; Self-complexity Measure; FSKN) | Pre-/ Post-Design, including 3 points of measurement: at the beginning of therapy/ waiting period; immediately after completion of therapy/ waiting period; catamnestic measurement 6 months later
Psychopathology/ Affect (ADS; PANAS) | Pre-/ Post-Design, including 3 points of measurement: at the beginning of therapy/ waiting period; immediately after completion of therapy/ waiting period; catamnestic measurement 6 months later
Community Integration (CIQ) | Pre-/ Post-Design, including 3 points of measurement: at the beginning of therapy/ waiting period; immediately after completion of therapy/ waiting period; catamnestic measurement 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Exner, Dr. (PhD), Principal Investigator — Philipps University Marburg, Department of Clinical Psychology and Psychotherapy; Winfried Rief, Prof. Dr., Study Director — Philipps University Marburg, Department of Clinical Psychology and Psychotherapy
Locations (2):
- Germany (2):
  - Philipps University Marburg, Departement of Clinical Psychology and Psychotherapy, Marburg
  - Psychotherapie-Ambulanz Marburg, Marburg

REFERENCES:
- See also: Click here for more information about this study: "Selbständig leben nach einer Hirnschädigung" — http://www.psychotherapie-ambulanz-marburg.de/FrameSets/fsForschung.html